CLINICAL TRIAL: NCT00958165
Title: Clinical Study of the CardioFocus Endoscopic Ablation System - Adaptive Contact (CFEAS- AC) for the Treatment of Symptomatic Atrial Fibrillation
Brief Title: Clinical Study of the CardioFocus Endoscopic Ablation System for the Treatment of Symptomatic AF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: CardioFocus (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-2738
Record Dates: First submitted 2009-08-12; First posted 2009-08-13 (Estimated); Results first posted 2016-07-27 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-07

CONDITIONS: Paroxysmal Atrial Fibrillation
Keywords: Treatment of PAF using EAS-AC
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- EAS-AC (Experimental): PVI with EAS-AC
  Interventions: Device: CardioFocus EAS-AC

INTERVENTIONS:
Device: CardioFocus EAS-AC — PVI for PAF

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of the endoscopic ablation system - adaptive contact (EAS-AC) in treated paroxysmal atrial fibrillation (PAF) with pulmonary vein isolation (PVI).

ELIGIBILITY:
Inclusion Criteria:

* Symptomatic, Paroxysmal atrial fibrillation (AF)
* 18 to 70 years of age
* Failure of at least one AAD
* Others

Exclusion Criteria:

* Generally good overall health as determined by multiple criteria
* Willing to participate in a study
* Others

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2009-08; Primary Completion 2012-03 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (3):
- Germany (3):
  - Cardioangiologisches Centrum Bethanien - CCB, Frankfurg
  - St. Georg Hosptial, Hamburg
  - Universität Leipzig - Herzzentrum, Leipzig

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EAS-AC
Started | 81 (81 enrolled participants resulted in 72 eligible participants that were treated.)
Treated | 72
Completed | 67 (Of the 72 treated participants, 67 completed follow-up and were evaluable for effectiveness.)
Not Completed | 14
Not completed — Lost to Follow-up | 5
Not completed — Not eligible | 9

BASELINE CHARACTERISTICS:
Population: Of the 81 enrolled participants, 72 meet all enrollment criteria and were treated. These are the evaluable baseline participants
Arm/Group | EAS-AC
Number analyzed (Participants) | 72
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34
  Male | 38
Region of Enrollment [Number; unit: participants]
  Germany | 72

OUTCOME MEASURES:

1. Primary Outcome: Chronic Effectiveness in Treating PAF as Demonstrated by no AF Recurrences After the Blanking Period and During the 12-month Follow-up Period.
Time Frame: 12 months
Population: Of the 72 enrolled and treated participants, 67 were evaluable for the chronic effectiveness endpoint.
Measure: Number; unit: Successful participants
Groups:
- EAS-AC: Pulmonary vein isolation treatment with EAS-AC for PAF
Arm/Group | EAS-AC
Number analyzed (Participants) | 67
Successful participants | 42

ADVERSE EVENTS:
Arm/Group | EAS-AC
Serious Adverse Events (participants affected / at risk) | 10/72
Other Adverse Events (participants affected / at risk) | 0/72
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | EAS-AC (N=72)
Phrenic nerve injury (Musculoskeletal and connective tissue disorders) | 1 (1)
Air embolism (Cardiac disorders) | 2 (2)
Pericardial tamponade (Cardiac disorders) | 4 (4)
Pericardial effusion (Cardiac disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No